CLINICAL TRIAL: NCT06521801
Title: Barts Health Cardio-Renal Registry
Brief Title: Cardio-Renal Registry
Acronym: BHCRR
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: BHCRR
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease; Cardio-Renal Syndrome; Myocardial Infarction; Cerebrovascular Accident; Percutaneous Coronary Intervention; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Cardio-Renal Syndrome; Myocardial Infarction; Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Renal Disease or Cardiology Disease: This study aims to assess, in a real-world setting, the safety, efficacy and feasibility of further investigations in patients with renal disease and cardiac disease.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
Cardiovascular disease is the leading cause of morbidity and mortality among patients with chronic kidney disease (CKD). Even after adjustment for known cardiovascular risk factors, including diabetes and hypertension, mortality risk progressively increases with worsening CKD. As glomerular filtration rate (GFR) declines the probability of developing coronary artery disease (CAD) increases linearly, and patients with GFR <60 mL/min/1.73 m2 have 2-3-fold increased CV mortality risk, relative to patients without CKD. Management of CAD is complicated in CKD patients due to the likelihood of comorbid conditions and potential for side effects. Despite their high cardiovascular risk, ACS patients with renal dysfunction are less commonly treated with guideline-based medical therapy and are less frequently referred for coronary revascularisation. This observation, referred to as the "treatment risk paradox," has been well described and may be explained by physicians' concerns regarding possible nonrenal side effects as well as renal toxicities. Furthermore, patients with severe CKD have traditionally been under-represented in most large cardiovascular clinical trials. Therefore, recommendations for both medical and revascularisation of CAD have relied heavily on extrapolation of results from the non-CKD population.

This data will add to that literature by assessing the characteristics and outcomes of patients with CAD and CKD. It will also identify and characterise predictors of outcomes, improve risk stratification and diagnostic evaluation.

ELIGIBILITY:
Informed consent will not be sought for, as patients are automatically included onto a database that we will use for research purposes. No children will be included in this study. Vulnerable adults or those unable to give consent will be included in the study as well if they are referred to the Nephrology team.

Inclusion Criteria:

1. Both male and female patients ≥16 years of age will be included
2. All patients will be reviewed by the Nephrology team a the RLH with renal disease.

Exclusion Criteria:

1. Patients <16 years will not be included in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients admitted to or reviewed at The Royal London Hospital (RLH) who have renal disease. These patients range from young adults to the elderly and will include any patient ≥16 years of age. Patients will include those who have end stage renal disease, seen in the low clearance clinic, are on dialysis, are on the renal transplant list and who are post renal transplant.
  Patients will be included from referrals made by other clinicians either as in or outpatients. All these patients have their clinical data captured on a database or hospital based clinical programme.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days and 1 year
Re-admission rates | 30 days and 1 year
Major Adverse Cardiac Events | 30 days and 1 year
Major Adverse Kidney Events | 30 days and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No